CLINICAL TRIAL: NCT04665895
Title: A Phase III, Randomized, Multicenter, Parallel-group Clinical Trial for Examining the Therapeutic Equivalence Between Fluticasone Propionate 100 mcg/Blister Oral Inhalation Powder/Respirent Pharmaceuticals vs. FLOVENT DISKUS® 100 mcg/Blister Oral Inhalation Powder/GSK in Patients With Asthma
Brief Title: A Clinical Trial for Examining the Therapeutic Equivalence Between Fluticasone Propionate 100 mcg/Blister Oral Inhalation Powder/Respirent Pharmaceuticals vs. FLOVENT DISKUS® 100mcg/Blister Oral Inhalation Powder/GSK in Patients With Asthma
Acronym: ANASSA-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Respirent Pharmaceuticals Co Ltd. (Industry)
Collaborators: Becro Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BECRO/RESP/ANASSA-PD
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Asthma
Keywords: asthma; therapeutic equivalence; bioequivalence; fluticasone propionate
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Test Product (Experimental): Fluticasone propionate 100 mcg/blister oral inhalation powder/Respirent Pharmaceuticals
  Interventions: Drug: Fluticasone propionate 100 mcg/blister oral inhalation powder/Respirent Pharmaceuticals
- Reference Product (Active Comparator): FLOVENT DISKUS® 100 mcg/blister oral inhalation powder/GSK
  Interventions: Drug: FLOVENT DISKUS® 100 mcg/blister oral inhalation powder/GSK
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate 100 mcg/blister oral inhalation powder/Respirent Pharmaceuticals — twice daily inhalation throughout the study
  Arms: Test Product
Drug: FLOVENT DISKUS® 100 mcg/blister oral inhalation powder/GSK — twice daily inhalation throughout the study
  Other Names: FLOVENT
  Arms: Reference Product
Drug: Placebo — twice daily inhalation throughout the study
  Arms: Placebo

SUMMARY:
Τherapeutic equivalence, randomized, multiple-dose, placebo-controlled, observer-blind, parallel group design consisting of a 2-week run-in period followed by a 4-week treatment period with Fluticasone propionate 100 mcg/ blister oral inhalation powder/Respirent Pharmaceuticals (Test) or FLOVENT DISKUS® 100mcg blister oral inhalation powder (Reference) or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects (≥12 years of age) of non-childbearing or of childbearing potential committed to consistent and correct use of an acceptable method of birth control.
2. Patients diagnosed with asthma, as defined by the National Asthma Education and Prevention Program (NAEPP), at least 12 weeks months prior to screening (Visit 1).
3. Pre-bronchodilator FEV1 of ≥45% and ≤85% of the predicted value (for age ≥18 years), or ≥65% and ≤90% predicted normal value (for ages 12 to 17 years) during the screening visit and on the first day of treatment.
4. Currently non-smoking; had not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and had ≤ 10 pack-years of historical use.
5. ≥12% and 200 mL reversibility of FEV1 within 30 minutes following 400 mcg salbutamol (4 puffs) inhalation (pMDI). This may be demonstrated at the Screening Visit or this test may be repeated on a different day if the patient fails the first attempt anytime in the period leading up to the day of randomization; If reversibility is not demonstrated up to the day of randomization then patients may be permitted to enter the study with historical evidence of reversibility that was performed within 2 years prior to Screening visit (Visit 1).
6. Patients should be on stable doses of their chronic asthma treatment regimen and should have well-controlled asthma for at least 4 weeks prior to enrolment.
7. Patients who are able to discontinue their asthma medications (inhaled corticosteroids and long-acting β agonists) during the run-in period and for the remainder of the study, according to investigator's judgement.
8. Patients who are able to replace current short-acting β agonists (SABAs) with salbutamol inhaler for use as needed for the duration of the study (subjects should be able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits).
9. Patients who are able to continue treatment with theophylline or montelukast without a significant adjustment of dosage, formulation, dosing interval for the duration of the study, and judged able by the investigator to withhold them for the specified minimum time intervals prior to each patient visit: 1) montelukast 36 hours 2) short-acting forms of theophylline 12 hours, 3) twice-a-day controlled-release forms of theophylline 24 hours, 4) once-a-day controlled-release forms of theophylline 36 hours.
10. Patients who are able to understand the requirements of the clinical trial and to agree to return for the required follow-up visits.
11. Willing to provide voluntary written informed consent and data protection declaration (and in the case of a minor their parent/guardian was able to give) before any clinical trial related procedure is performed.

Exclusion Criteria:

1. Life-threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnia; respiratory arrest or hypoxic seizures, asthma related syncopal episode(s), or hospitalizations within the past year.
2. Significant respiratory disease other than asthma (COPD, interstitial lung disease, chronic bronchitis, emphysema, etc.).
3. Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic neurologic, psychiatric, renal, or other diseases that in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
4. Hypersensitivity to any sympathomimetic drug (e.g. salbutamol) or any inhaled, intranasal, or systemic corticosteroid therapy.
5. History of hypersensitivity to lactose.
6. Patients receiving β-blockers, anti-arrhythmics, polycyclic antidepressants and/or monoamine oxidase inhibitors within 4 weeks prior to the screening.
7. Asthma exacerbation (i.e. acute or sub-acute worsening in symptoms and lung function from the patient's usual status) or symptoms or signs of viral or bacterial, upper or lower respiratory tract infection or sinus or middle ear infection within 4 weeks prior to the screening visit or during the run-in period.
8. Use of oral or parenteral corticosteroids within 12 weeks prior to Screening visit (Visit 1)
9. Factors (e.g., infirmity, disability or geographic location) that the investigator felt would likely limit the patient's compliance with the study protocol or scheduled clinic visits.
10. Female Subjects who are pregnant or breastfeeding.
11. Women of child-bearing age that are not surgically incapable of pregnancy and are not willing to use an acceptable method of birth control.
12. Current participation or not yet completed period of at least 30 days since ending other investigational device or drug trial(s).
13. Unwillingness or inability to comply with the clinical trial procedures;
14. Unwillingness to consent to storage, saving and transmission of pseudonymous medical data for clinical trial reasons;
15. Who are legally incapacitated;
16. Who are legally detained in an official institute

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Pre-dose FEV1 | 28-days
  FEV1 measured in the morning prior to the dosing of inhaled medications on the last day of a 28-days treatment after adjustment for baseline

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Kostikas, Associate Professor, Principal Investigator — University of Ioannina Department of Medicine
Locations (1):
- BECRO Ltd., Athens, Greece

IPD SHARING:
Plan to Share IPD: No